CLINICAL TRIAL: NCT03235115
Title: Fitting Evaluation of Hydrogel and Silicone Hydrogel Spherical Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-85
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Results first posted 2018-11-14 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Methafilcon A IV (Active Comparator): Subjects are randomized to wear Methafilcon A IV for 1 hour during the cross over study.
  Interventions: Device: Ocufilcon B; Device: Omafilcon A
- Ocufilcon B (Active Comparator): Subjects are randomized to wear Ocufilcon B for 1 hour during the cross over study.
  Interventions: Device: Methafilcon A IV; Device: Omafilcon A
- Omafilcon A (Active Comparator): Subjects are randomized to wear Omafilcon A for 1 hour during the cross over study.
  Interventions: Device: Methafilcon A IV; Device: Ocufilcon B

INTERVENTIONS:
Device: Methafilcon A IV — Contact Lens
  Arms: Ocufilcon B; Omafilcon A
Device: Ocufilcon B — Contact Lens
  Arms: Methafilcon A IV; Omafilcon A
Device: Omafilcon A — Contact Lens
  Arms: Methafilcon A IV; Ocufilcon B

SUMMARY:
This study aims to compare the short-term clinical performance of the three contact lenses (Methafilcon A IV, Ocufilcon B 1-day and Omafilcon A 1-day daily disposable).

DETAILED DESCRIPTION:
This will be a randomized, double-masked, crossover, bilateral non-dispensing study, controlled by cross-comparison. Forty subjects will wear each lens brand for approximately one hour, on three separate study days in random order. Lenses will only be worn during study visits.

ELIGIBILITY:
Inclusion Criteria:

* They are of aged 18-40 and have capacity to volunteer.
* They understand their rights as a research subject and are willing and able to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They agree not to participate in other clinical research for the duration of this study.
* They have a contact lens spherical prescription between -1.00 to - 6.00D (inclusive)
* They have a spectacle cylindrical correction of -0.75D or less in each eye (based on the ocular refraction).
* They can attain at least 0.10 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
* They currently use soft contact lenses or have done so in the previous six months.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They have had cataract surgery.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
* They are pregnant or lactating.
* They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear.
* They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
* They have taken part in any other contact lens or care solution clinical trial or research, within two weeks prior to starting this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research - The University of Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Methafilcon A IV, Ocufilcon B, Omafilcon A: Subjects randomized to wear Methafilcon A IV first, then Ocufilcon B, then Omafilcon A contact lens
- Methafilcon A IV, Omafilcon A, Ocufilcon B: Subjects randomized to wear Methafilcon A IV first, then Omafilcon A, then Ocufilcon B contact lens
- Ocufilcon B, Omafilcon A, Methafilcon A IV: Subjects randomized to wear Ocufilcon B first, then Omafilcon A, then Methafilcon A IV contact lens
- Ocufilcon B, Methafilcon A IV, Omafilcon A: Subjects randomized to wear Ocufilcon B first, then Methafilcon A IV, then Omafilcon A contact lens
- Omafilcon A, Ocufilcon B, Methafilcon A IV: Subjects randomized to wear Omafilcon A first, then Ocufilcon B, then Methafilcon A IV contact lens
- Omafilcon A, Methafilcon A IV, Ocufilcon B: Subjects randomized to wear Omafilcon A first, then Methafilcon A IV, then Ocufilcon B contact lens
Period: First Intervention (1 Hour, Visit 2)
Arm/Group | Methafilcon A IV, Ocufilcon B, Omafilcon A | Methafilcon A IV, Omafilcon A, Ocufilcon B | Ocufilcon B, Omafilcon A, Methafilcon A IV | Ocufilcon B, Methafilcon A IV, Omafilcon A | Omafilcon A, Ocufilcon B, Methafilcon A IV | Omafilcon A, Methafilcon A IV, Ocufilcon B
Started | 9 | 6 | 7 | 6 | 6 | 6
Completed | 9 | 6 | 7 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Period: Second Intervention (1 Hour, Visit 4)
Arm/Group | Methafilcon A IV, Ocufilcon B, Omafilcon A | Methafilcon A IV, Omafilcon A, Ocufilcon B | Ocufilcon B, Omafilcon A, Methafilcon A IV | Ocufilcon B, Methafilcon A IV, Omafilcon A | Omafilcon A, Ocufilcon B, Methafilcon A IV | Omafilcon A, Methafilcon A IV, Ocufilcon B
Started | 9 | 6 | 7 | 6 | 6 | 5
Completed | 9 | 6 | 7 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention ( 1 Hour, Visit 6)
Arm/Group | Methafilcon A IV, Ocufilcon B, Omafilcon A | Methafilcon A IV, Omafilcon A, Ocufilcon B | Ocufilcon B, Omafilcon A, Methafilcon A IV | Ocufilcon B, Methafilcon A IV, Omafilcon A | Omafilcon A, Ocufilcon B, Methafilcon A IV | Omafilcon A, Methafilcon A IV, Ocufilcon B
Started | 9 | 6 | 7 | 6 | 6 | 5
Completed | 9 | 6 | 7 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants were randomized to wear each of the 3 different contact lens pairs
Arm/Group | All Study Participants
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Using logMAR
Description: Assessment of visual performance using the Bailey-Lovie logMAR visual acuity test chart and procedures for carrying out an over-refraction
Time Frame: Dispense and follow-up, approximately one hour (1hr) of lens wear for each lens type worn
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Omafilcon A: Subjects who wore Omafilcon A for 1 hour during the cross over study.
- Methafilcon A IV: Subjects who wore Methafilcon A IV for 1 hour as one of the 3 lenses in this crossover study.
- Ocufilcon B: Subjects who wore Ocufilcon B for 1 hour as one of the 3 lenses in this crossover study.
Arm/Group | Omafilcon A | Methafilcon A IV | Ocufilcon B
Number analyzed (Participants) | 40 | 39 | 39
logMAR
  At Dispense | -0.14 (0.09) | -0.13 (0.07) | -0.13 (0.07)
  Follow Up | -0.14 (0.07) | -0.14 (0.07) | -0.14 (0.07)

2. Primary Outcome: Lens Fit - Horizontal Centration
Description: Assessment of horizontal centration of lens on eye
Time Frame: Dispense and follow-up, approximately one hour (1hr) of lens wear for each lens type worn
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Methafilcon A IV | Ocufilcon B
Number analyzed (Participants) | 40 | 39 | 39
Participants
  At dispense: Extremely nasal | 0 | 0 | 0
  At dispense: Slightly nasal | 1 | 1 | 1
  At dispense: Optimum | 23 | 17 | 26
  At dispense: Slightly temporal | 16 | 21 | 12
  At dispense: Extremely temporal | 0 | 0 | 0
  At follow up: Extremely nasal | 0 | 0 | 0
  At follow up: Slightly nasal | 1 | 2 | 0
  At follow up: Optimum | 22 | 14 | 26
  At follow up: Slightly temporal | 17 | 22 | 13
  At follow up: Extremely temporal | 0 | 1 | 0

3. Primary Outcome: Lens Fit - Vertical Centration
Description: Assessment of vertical centration of lens on eye
Time Frame: Dispense and follow-up, approximately one hour (1hr) of lens wear for each lens type worn
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Methafilcon A IV | Ocufilcon B
Number analyzed (Participants) | 40 | 39 | 39
Participants
  At dispense: Extremely inferior | 0 | 0 | 0
  At dispense: Slightly inferior | 12 | 6 | 9
  At dispense: Optimum | 20 | 9 | 27
  At dispense: Slightly superior | 8 | 24 | 3
  At dispense: Extremely superior | 0 | 0 | 0
  At follow up: Extremely inferior | 0 | 0 | 0
  At follow up: Slightly inferior | 15 | 4 | 11
  At follow up: Optimum | 18 | 14 | 26
  At follow up: Slightly superior | 7 | 21 | 2
  At follow up: Extremely superior | 0 | 0 | 0

4. Primary Outcome: Lens Fit - Corneal Coverage of Lens
Description: Assessment of corneal coverage of lens on eye
Time Frame: Dispense and follow-up, approximately one hour (1hr) of lens wear for each lens type worn
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Methafilcon A IV | Ocufilcon B
Number analyzed (Participants) | 40 | 39 | 39
Participants
  At dispense: Extremely inadequate | 0 | 0 | 0
  At dispense: Slightly inadequate | 6 | 16 | 4
  At dispense: Optimum | 29 | 22 | 30
  At dispense: Slightly excessive | 5 | 1 | 5
  At dispense: Extremely excessive | 0 | 0 | 0
  At follow up: Extremely inadequate | 0 | 1 | 0
  At follow up: Slightly inadequate | 5 | 13 | 4
  At follow up: Optimum | 30 | 24 | 30
  At follow up: Slightly excessive | 5 | 1 | 5
  At follow up: Extremely excessive | 0 | 0 | 0

5. Primary Outcome: Lens Fit - Movement of Lens
Description: Assessment of movement of lens on eye
Time Frame: Dispense and follow-up, approximately one hour (1hr) of lens wear for each lens type worn
Measure: Count of Participants; unit: Participants
Arm/Group | Omafilcon A | Methafilcon A IV | Ocufilcon B
Number analyzed (Participants) | 40 | 39 | 39
Participants
  At dispense: Extremely inadequate | 0 | 0 | 0
  At dispense: Slightly inadequate | 1 | 7 | 8
  At dispense: Optimum | 24 | 25 | 16
  At dispense: Slightly excessive | 15 | 7 | 15
  At dispense: Extremely excessive | 0 | 0 | 0
  At follow up: Extremely inadequate | 0 | 0 | 0
  At follow up: Slightly inadequate | 2 | 2 | 1
  At follow up: Optimum | 23 | 28 | 19
  At follow up: Slightly excessive | 15 | 9 | 19
  At follow up: Extremely excessive | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Patients wore 3 different contact lenses for 1 hour on 3 different days
Arm/Group | Omafilcon A | Methafilcon A IV | Ocufilcon B
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/39
Other Adverse Events (participants affected / at risk) | 0/40 | 0/39 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restriction on the PI is that the sponsor should be notified of any use of data for results communication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT03235115/Prot_SAP_001.pdf